CLINICAL TRIAL: NCT00055978
Title: Lung Cancer Chemoprevention With Celecoxib In Ex-Smokers
Brief Title: Celecoxib in Preventing Lung Cancer in Former Heavy Smokers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Jenny T. Mao, Jonsson Comprehensive Cancer Center at UCLA
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CDR0000271912; U01CA096134 (NIH); P30CA016042 (NIH); UCLA-0108074
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2011-06

CONDITIONS: Lung Cancer
Keywords: non-small cell lung cancer; stage I non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive oral placebo twice daily for 6 months.
  Interventions: Other: placebo
- Arm II (Experimental): Patients receive oral celecoxib twice daily for 6 months.
  Interventions: Drug: celecoxib

INTERVENTIONS:
Drug: celecoxib — Given orally. 400mg twice daily for 6 months.
  Other Names: Celebrex; Celebra
  Arms: Arm II
Other: placebo — Given orally
  Arms: Arm I

SUMMARY:
RATIONALE: Chemoprevention therapy uses certain drugs to try to prevent the development or recurrence of cancer. Celecoxib may be effective in preventing the development or recurrence of lung cancer in former heavy smokers.

PURPOSE: Randomized phase II trial to study the effectiveness of celecoxib in preventing the development or recurrence of lung cancer in former heavy smokers who are at risk of developing cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of chemoprevention of lung cancer with celecoxib in former heavy smokers at risk for developing primary or second primary lung cancer.
* Determine the safety and side effects of this drug in these patients.
* Determine the quality of life of patients treated with this drug.
* Determine the role of COX-2-specific inhibitors (e.g., celecoxib) on antitumor immunity within the lung microenvironment of these patients.
* Determine the effects of COX-2 inhibition on angiogenesis in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are stratified according to presence of preinvasive lesions (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral placebo twice daily for 6 months.
* Arm II: Patients receive oral celecoxib twice daily for 6 months. Treatment in both arms continues in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed every 6 months during treatment and then annually for up to 4 years.

Patients are followed annually for up to 4 years.

PROJECTED ACCRUAL: A total of 180 patients (90 per treatment arm) will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Heavy former smokers without prior history of NSCLC

  * Age > 45
  * Smoked for minimum of 30 pack years
* Former smokers with prior curative resection of surgical stage I NSCLC will be recruited and must be:

  * Age > 18
  * Smoked > 10 pack years
  * Must have had pathological staging and the extent of disease documented. At least one nodal station each must have been biopsied and all biopsies must have been negative
  * At least 6 months post curative resection of Stage I prior NSCLC, without evidence for recurrence or second primary lung cancer
* Normal blood chemistry and cell counts
* Negative pregnancy test

Exclusion Criteria:

* Framingham 10-year-risk for coronary artery disease score > 10%
* History of cardiovascular disease
* Evidence of diffuse coronary calcification on screening CT
* Concurrent use of NSAIDs. The use of cardiac (baby) Aspirin is permitted
* Hypersensitivity to celecoxib, sulfonamides, aspirin or other NSAIDs
* Liver dysfunction [abnormally elevated liver function tests [transaminases (ALT, AST) > ULN, alkaline phosphatase (ALKP) > 1.5 ULN]] or history of cirrhosis
* No peptic ulcer disease (PUD) diagnosis nor active symptoms in the last 2 years or, if PUD was diagnosed < 2 years, there must be no active symptoms, and endoscopic confirmation of healing
* Renal dysfunction [abnormally elevated blood urea nitrogen (BUN) > 1.5 ULN and creatinine > ULN]
* End state respiratory disease
* Unstable angina or a history of significant coronary artery disease
* Other malignancies excluding non-melanoma type skin cancer and in situ cervical cancer. Persons with stage I/II head and neck cancer must be disease free for at least 12 months
* Pregnancy
* Lactation
* Unwillingness to practice contraception
* On systemic corticoid steroid therapy
* Coagulopathy
* Use of Coumadin
* Concurrent use of medication know to alter or be affected by alteration of hepatic p450 2C9 enzymes.
* Patients with concurrent medical conditions that may interfere with completion of tests, therapy, or the follow up schedule
* Patients who had received photosensitizing agents such as hematoporphyrin derivative or chemopreventive drugs such as retinoids within 3 months prior to the bronchoscopic procedure, radiotherapy to the chest, or cytotoxic chemotherapy agents
* Subject found to have CIS during screening bronchoscopy will be treated with local therapy prior to randomization

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2002-10; Primary Completion 2008-03 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Modulation of the ki-67 labeling index | 5 years
Phenotypic modulation of the bronchial histology | 5 years

SECONDARY OUTCOMES:
Evidence of molecular/genetic aberrations | 5 years
Changes indicative of response to treatment in the targeted signaling pathway | 5 years
Parameters that reflect the overall balance of the epigenetic phenomenon thought to facilitate or promote tumorigenesis | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jenny T. Mao, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States